CLINICAL TRIAL: NCT00785304
Title: ADVANCED MRI IN BLAST-RELATED TBI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Washington University School of Medicine (Other)
Collaborators: Landstuhl Regional Medical Center (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Brody, MD, PhD, Associate Professor of Neurology, Washington University School of Medicine
Other Study IDs: PT075299
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Traumatic Brain Injury: Active Duty military blast-related TBI patients
- Other Injury Control: Active duty military patients with other injuries but no TBI

SUMMARY:
Thousands of soldiers, marines, and other military personnel have had injuries to the brain due the wars in Iraq and Afghanistan. In addition, 1.5 million civilians per year in the United States have traumatic brain injuries caused by car accidents, falls, sports-related injuries or assaults. There are important advances in technology that we think will help us learn a lot more about these injuries. One such advance involves new types of MRI scans that we think will be able to show what has happened to the brain after trauma more clearly that regular scans can. These first new scan is called diffusion tensor imaging, which shows injury to the axons (the wiring of the brain). The second new scan is called resting-state functional MRI correlation analysis, which shows how well various parts of the brain are connected to each other. Importantly, the new types of scans can be done using regular scanners that we already have in every major hospital. The innovation is entirely in how the scanners are used and how the resulting pictures are analyzed on a computer after they have been taken.

Our overall goal is to see whether these new MRI scans will be useful for people who have had traumatic brain injuries. We have already tested them on some civilian brain injury patients and found them to be very helpful. For this study, we will test them on military personnel who have had traumatic brain injuries caused by explosions. The specific goal will be to see if the amount of injury we see can be used to predict how well the patients will do overall over the next 6-12 months. We think with the new scans we will be able to predict overall outcomes better than with regular scans and other information. A related goal will be to see whether injuries to specific parts of the brain seen by these new scans can be used to predict whether patients will be likely to have specific problems like memory loss, attention deficit, depression, or post-traumatic stress disorder. A final goal will be to repeat the scans 6-12 months later to see whether the new MRI scans can show whether the injuries to the brain have healed, gotten worse, or stayed the same.

If the study is successful, it will show that these new MRI techniques can to be used to make earlier and more accurate diagnoses of traumatic brain injury, predictions of the sorts of problems that are likely to occur after brain injury, and assessments of how severe the injuries are.

This study will help traumatic brain injury patients. It will be most useful for military personnel who have had brain injuries due to explosions. It is highly likely that it will also be useful for younger adults who have had brain injuries due to other causes like car accidents, sports-related concussions, falls, or assaults. It is possible that but not known for sure whether it will help young children or older adults with traumatic brain injuries.

These new scans could help with decisions about whether military personnel can return to duty, what sort of rehabilitation would benefit them most, and what family members should watch for and expect. This could become used in some hospitals within 2 years, and could become standard in every major hospital within 5 years.

The new scans could also be helpful in developing new treatments. For example, if a new drug works by blocking injury to the axons, it would be a good idea to test on people who have injury to their axons. Right now we have no good way to tell who these people are, and so a new drug like this would get tested on lots of people who don't have injured axons, along with those who do. This would make it harder to tell if the new drug is working. With the new scans we should be able to tell who has injured axons, tell how severe the injury is, and figure out whom to test the drugs on. It will likely take 10 years or more to develop new drugs like this.

Further in the future, the new scans could be used to help guide surgery to implant computer chips to help rewire the brain. We don't know how long this will take, but estimate 15-20 years or more.

Overall MRI scanning is very safe and has no known major risks. Because the scanner uses strong magnets, anyone with metal objects in their bodies can't be scanned, as this could be dangerous. We will make sure that no one with metal objects in their bodies is included in the study. There can be some psychological risks involved in taking tests and answering questions, but these are usually mild and can be managed. There is always a risk that important confidential information will be made public and that this could have consequences. We will do everything possible to maintain confidentiality. Nearly all of the information will only be identified using a code number and not by the name of the person, and all of it will be kept securely.

DETAILED DESCRIPTION:
Background: In traumatic brain injury, axonal damage is a major pathophysiological process and may be a primary cause of adverse neurological outcomes. However, traumatic axonal injury and its effects on brain functional connectivity are very difficult to directly detect and quantify in living patients. Diffusion tensor imaging (DTI) appears to have great promise with regard to detecting axonal injury. Resting-state fMRI correlation analysis likewise may be a powerful and broadly applicable method for investigating brain functional connectivity. In our preliminary studies, these two techniques have been successfully used together in several civilian TBI patients. They appear to synergistically cross validate each other; disrupted functional connectivity underlying focal neurological deficits were revealed using resting-state fMRI correlation analysis while DTI demonstrated the axonal injury responsible for the disruptions. Conventional MRI and CT entirely failed to explain many of these deficits. This cross validation is important as it adds confidence to the interpretation of the results. Without resting-state fMRI correlation analysis, the consequences of apparent axonal injury on DTI for the functional connectivity of the brain may not be clear; the axonal injury could be in white matter tracts that are redundant, or not severe enough to be functionally important. Without DTI, the cause of a disruption in connectivity seen using resting-state fMRI correlation analysis will likewise not always be known; processes other than traumatic axonal injury could be responsible. Both of these advanced techniques along with a full conventional MRI can be performed on standard clinical MRI scanners in approximately 45 minutes per patient. Apart from in our preliminary studies, resting-state fMRI and DTI have not been used together to investigate traumatic brain injury.

Objective/Hypothesis: The objective of this proposal is to test these two advanced MRI methods, DTI and resting-state fMRI, in active-duty military blast-related TBI patients acutely after injury and correlate findings with TBI-related clinical outcomes 6-12 months later. These methods may add clinically useful predictive information following traumatic brain injury that could be of assistance in standardizing diagnostic criteria for TBI, making return-to-duty triage decisions, guiding post-injury rehabilitation, and developing novel therapeutics. The overarching hypothesis guiding this project is that traumatic axonal injury is a principal cause of impaired brain function following blast-related TBI. Specific hypotheses to be tested are:

1. DTI and resting-state fMRI correlation analysis will noninvasively reveal abnormalities that are not present on CT or conventional MRI acutely following blast-related TBI.
2. Specific patterns of acute axonal injury (on DTI) causing disruption of brain functional connectivity (on resting-state fMRI correlation analysis) will predict specific neurological, neuropsychological, and psychiatric deficits and disorders.
3. The overall burden of acute axonal injury and disrupted brain functional connectivity will strongly predict overall 6-12 month clinical outcome.

Specific Aims: 1) to obtain DTI, resting-state fMRI and conventional MRI scans acutely after blast-related TBI in active-duty military personnel presenting to Landstuhl Regional Medical Center (LRMC).

2) to collect detailed clinical information on TBI-related outcomes 6-12 months after injuries.

3) to extensively analyze the acute imaging predictors and correlates of 6-12 month clinical outcomes.

Study Design: We propose a prospective, observational study of 80 active duty military personnel who have sustained blast-related TBI. Initial scans will be performed within 4 days of injury at LRMC. Follow-up will occur monthly by telephone and in person at Washington University 6-12 months after injury. Clinical information on TBI outcomes collected will include global outcome assessments, neuropsychological testing for memory, attention and executive function deficits, motor performance measures, and clinician administered rating scales for depression and post-traumatic stress disorder. Controls will include 1) an additional group of 20 active duty military personnel with other injuries, but who have not had TBI, and 2) age, gender and education-based norms for standardized test and assessment results. Repeat DTI, resting-state fMRI, and conventional MRI will be performed to track the evolution of the injuries. Analysis approaches will include prespecified hypotheses based on known brain anatomical-clinical correlations and several exploratory approaches, as the structural bases for many post-traumatic neurological and neuropsychological deficits are not well understood. Non-parametric correlational statistical methods and rigorous correction for multiple comparisons will be employed. Expert collaborators and logistics coordinators will be or have already been recruited. Confidentiality and privacy will be tightly controlled.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of blast-related TBI of any severity, as made by LRMC staff, based on clinical history, examination, and/or standard clinical imaging (CT, conventional MRI).
2. Acute injury or injuries, defined as first occurring 0-90 days prior to enrollment.
3. Ability to lie still in a supine position for the duration of the scan sessions, e.g. no severe claustrophobia or limiting pain from other injuries.
4. No known metallic implants or metallic foreign objects.
5. Ability to provide informed consent.
6. Not known to be HIV positive
7. Not known to be pregnant
8. No previous major traumatic brain injury
9. No contraindication to MRI for medical reasons such as arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active duty military personnel serving in Iraq, Afghanistan, and other areas presenting to Landstuhl Regional Medical Center for care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of the overall extent of abnormalities apparent on DTI vs conventional MRI. | 1 year
Identification of specific injured white matter tracts. | 1 year
Assessment of the correlations in fMRI signal fluctuations between brain regions. | 1 year
Prediction of the 6-12 month global clinical outcome (GOS-E) based on the acutely apparent DTI abnormalities. | 1 year
Prediction of the 6-12 month global clinical outcome (GOS-E) based on the acutely apparent resting fMRI correlation abnormalities. | 1 year
Prediction of the presence and clinical severity of specific post-traumatic sequelae, including i. Spastic hemi/tetraparesis:ii. Short-term learning and memory deficits:iii. Attention deficit:iv. Depression:v. Post-traumatic stress disorder: | 1 year
Comparison of acute and 6-12 month scans. | 1 year
Evaluation of the predictive value of the Military Acute Concussion Evaluation (MACE) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David L Brody, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (2):
- Washington University, St Louis, Missouri, United States
- Landstuhl Regional Medical Center, Landstuhl, Kirchberg, Germany

REFERENCES:
- [Result] Mac Donald CL, Johnson AM, Cooper D, Nelson EC, Werner NJ, Shimony JS, Snyder AZ, Raichle ME, Witherow JR, Fang R, Flaherty SF, Brody DL. Detection of blast-related traumatic brain injury in U.S. military personnel. N Engl J Med. 2011 Jun 2;364(22):2091-100. doi: 10.1056/NEJMoa1008069. PMID 21631321
- [Result] Mac Donald C, Johnson A, Cooper D, Malone T, Sorrell J, Shimony J, Parsons M, Snyder A, Raichle M, Fang R, Flaherty S, Russell M, Brody DL. Cerebellar white matter abnormalities following primary blast injury in US military personnel. PLoS One. 2013;8(2):e55823. doi: 10.1371/journal.pone.0055823. Epub 2013 Feb 7. PMID 23409052
- [Result] Han K, Mac Donald CL, Johnson AM, Barnes Y, Wierzechowski L, Zonies D, Oh J, Flaherty S, Fang R, Raichle ME, Brody DL. Disrupted modular organization of resting-state cortical functional connectivity in U.S. military personnel following concussive 'mild' blast-related traumatic brain injury. Neuroimage. 2014 Jan 1;84:76-96. doi: 10.1016/j.neuroimage.2013.08.017. Epub 2013 Aug 20. PMID 23968735
- [Result] MacDonald CL, Johnson AM, Nelson EC, Werner NJ, Fang R, Flaherty SF, Brody DL. Functional status after blast-plus-impact complex concussive traumatic brain injury in evacuated United States military personnel. J Neurotrauma. 2014 May 15;31(10):889-98. doi: 10.1089/neu.2013.3173. Epub 2014 Feb 10. PMID 24367929